CLINICAL TRIAL: NCT05701631
Title: Radiomics Model for the Diagnosis of Pneumocystis Jirovecii Pneumonia in Non-HIV Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Liang_An, Professor, Chinese PLA General Hospital
Other Study IDs: S2023-006-01
Record Dates: First submitted 2023-01-17; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Pneumocystis Jirovecii Pneumonia
Keywords: Computed tomography; Diagnostic tests; Pneumocystis jirovecii pneumonia; Radiomics
MeSH Terms: conditions — Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- non-HIV patients hospitalized for suspected PCP: non-HIV patients hospitalized for suspected PCP
  Interventions: Diagnostic Test: Radiomic model

INTERVENTIONS:
Diagnostic Test: Radiomic model — Radiomic model for PCP diagnosis

SUMMARY:
To evaluate the performance of radiomics in differentiating Pneumocystis jirovecii pneumonia (PCP) from other types of pneumonia and to improve the diagnostic efficacy of non-invasive tests in non-HIV patients.

DETAILED DESCRIPTION:
Retrospective study, including non-HIV patients hospitalized for suspected PCP from January 2010 to December 2022. The included patients were randomized in a 7:3 ratio into training and validation cohorts. Radiomic features were extracted from semi-automatically identified infected areas in computed tomography (CT) scans and used to construct a radiomic model, which was then compared to a clinical-imaging model built with clinical and semantic CT features in terms of diagnostic performance of PCP. The combination of the radiomic model and serum β-D-glucan levels was also evaluated for PCP diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* aged over eighteen years;
* presence of an underlying disease known to be associated with PCP
* symptoms of lower respiratory tract infection, such as fever, cough or dyspnea
* signs of lung infection on high resolution CT at the on-set of the disease
* received BAL examination within three days after CT scans
* underwent qPCR and IF staining tests on the BAL fluid sample.

Exclusion Criteria:

* with HIV infection
* taking trimethoprim-sulfamethoxazole for prophylaxis
* undiagnosed by qPCR and IF staining tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to our institute with clinical suspected PCP
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
the diagnostic performance of radiomic model in the PCP diagnosis | 6 months
  The included patients were randomized in a 7:3 ratio into training and validation cohorts. Radiomic features were extracted from semi-automatically identified infected areas in computed tomography (CT) scans and used to construct a radiomic model. Then, the area under the curve (AUC) of the receiver operating characteristic (ROC) curves were calculated and used to evaluate the diagnostic performance (accuracy, sensitivity, specialty, positive predictive value, negative predictive value) of the model for PCP diagnosis in both training and validation cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-an Chen, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Contact the researcher for requests.

REFERENCES:
- [Derived] Yu H, Yang Z, Wei Y, Shi W, Zhu M, Liu L, Wang M, Wang Y, Zhu Q, Liang Z, Zhao W, Chen LA. Computed tomography-based radiomics improves non-invasive diagnosis of Pneumocystis jirovecii pneumonia in non-HIV patients: a retrospective study. BMC Pulm Med. 2024 Jan 2;24(1):11. doi: 10.1186/s12890-023-02827-4. PMID 38167022